CLINICAL TRIAL: NCT05697263
Title: The Impact of the Menstrual Cycle on Physical Exercise and Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Angelica Hirschberg Lindén, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-01650
Record Dates: First submitted 2022-11-20; First posted 2023-01-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Menstrual Cycle; Exercise; Women's Health; Athletic Performance
Keywords: Menstrual Cycle; Exercise; Women's Health; Athletic Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The testleader will be blinded to which group the subject belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Follicle phase based training (Experimental): Follicular phase-based training five times a week during the follicular phase (the first two weeks of the menstrual cycle) and thereafter once a week for the rest of the cycle.
  Interventions: Other: Periodization of training
- Luteal phase based training (Experimental): Luteal phase-based training five times a week during the luteal phase (from ovulation to next menstruation) and once a week in the follicular phase.
  Interventions: Other: Periodization of training
- Regular training (Experimental): Regular training three times a week throughout the menstrual cycle (control group).
  Interventions: Other: Periodization of training

INTERVENTIONS:
Other: Periodization of training — Participants in the three arms will exercise the same dose and number of sessions distributed in three different ways.

SUMMARY:
The menstrual cycle implies a basic difference in the biology of women and men but the effect of the hormonal variation on training protocols and physical performance is still not fully understood. Despite no existing evidence, the advice to periodize exercise according to the menstrual cycle has been widely spread among elite athletes, coaches, and sports federations. The advice is based on underpowered studies with considerable methodological weaknesses regarding determination of cycle phase, inclusion of athletes and lack of adequate control groups.

The purpose of this randomized, controlled study is to evaluate the effect of exercise periodization on aerobic fitness during different phases of the menstrual cycle. Further, the effect will be related to premenstrual symptoms, body composition and skeletal muscle morphology, sex hormone receptors, metabolic enzymes, and markers of muscle protein synthesis. This study will be well controlled and follow methodology recommendations for menstrual cycle research in sports and exercise.

Female athletes of fertile age will be randomized to different training regimens during three menstrual cycles (12 weeks):

Group A: Training three times a week throughout the menstrual cycle. Group B: Follicular phase-based training five times a week during the follicular phase and thereafter once a week during the luteal phase.

Group C: Luteal phase-based training five times a week during the luteal phase and once a week in the follicular phase.

The exercise will consist of high intensity intermittent spinning classes. Assessment of aerobic fitness and power will be performed at baseline, and again after three completed menstrual cycles. On the same day, body composition will be examined by DXA and blood samples will be collected for analysis of hormones and binding proteins. To confirm menstrual cycle phase, blood samples will be collected for hormone determination, and urinary stick will be used for detection of ovulation. Subjective ratings of menstrual cycle related symptoms will be performed every day. In a subgroup of women, muscle biopsies will be collected from m vastus lateralis at baseline and at the end of the study. This study will contribute to improved knowledge about exercise periodization in relation to the menstrual cycle. Well-grounded data is crucial to give evidence-based recommendations to female athletes when planning their training protocol to optimize training results and performance.

ELIGIBILITY:
Inclusion Criteria:

* Women exercising at least 3-4 times a week on a high level
* Regular menstrual cycle with 26-32 cycle days.
* Fully healthy and be able to follow the training program.

Exclusion Criteria:

* Hormonal contraceptive users,
* Users of regular medication
* Chronic disease
* Past or present neurological disorder
* Recent musculoskeletal injury

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in aerobic performance | Change from baseline aerobic performance at the end of Cycle 4 (each cycle is around 28 days)
  Cosmeds K5 Wearable Metabolic System will be used for breath-by-breath gas exchange measurements. Change in VO2peak from baseline to end of study will be evaluated.

SECONDARY OUTCOMES:
Change in muscle strength | Change from baseline muscle strength at the end of Cycle 4 (each cycle is around 28 days)
  A standardized isokinetic device (Biodex®, Corp, Shirley, NY, USA) will be used for measurements of maximal muscle torque (Nm) in the leg extensor muscles at 90 and 120 gr/sec (11). Change in muscle strength from baseline to end of study will be compared between groups.
Change in one-leg sit-to-stand test | Change from baseline test at the end of Cycle 4 (each cycle is around 28 days)
  Assessment of functional muscle strength in the lower extremities.
Change in one-leg hop test for distance | Change from baseline test at the end of Cycle 4 (each cycle is around 28 days)
  Assessment of functional muscle strength in the lower extremities.
Change in body composition | Change from baseline body composition at the end of Cycle 4 (each cycle is around 28 days)
  Differences in body fat (%) will be determined by DXA (Lunar equipment).
Change in body composition | Change from baseline body composition at the end of Cycle 4 (each cycle is around 28 days)
  Differences in muscle mass (g), will be determined by DXA (Lunar equipment).
Premenstrual symptoms | Every day during the study period
  Prospective ratings of premenstrual symptoms will be performed with the Cyclicity Diagnoser
Change in metabolic serum markers | Change from baseline metabolic serum markers at the end of Cycle 4 (each cycle is around 28 days)
  Blood samples for analysis of IGF-1.
Change in mucle morphology | Change from baseline muscle morphology at the end of Cycle 4 (each cycle is around 28 days)
  Muscle biopsy in mm vastus lateralis
Change in muscle tissue steroid hormones | Change from baseline muscle tissue steroid hormones at the end of Cycle 4 (each cycle is around 28 days)
  Muscle biopsy in mm vastus lateralis
Change in muscle protein synthesis | Change from baseline muscle protein synthesis at the end of Cycle 4 (each cycle is around 28 days)
  Muscle biopsy in mm vastus lateralis
Dysmenorrhea | Through study completion, an average of 4 month
  Questionnaire

OTHER OUTCOMES:
Confirmation of menstrual cycle phase | Through study completion, an average of 4 months
  Blood sampels will be collected at early follicular phase, ovulation phase and mid luteal phase for analysis of LH, FSH, estradiol and progesterone.

CONTACTS AND LOCATIONS:
Locations (1):
- Angelica Lindén Hirschberg, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] von Rosen P, Ekenros L, Solli GS, Sandbakk O, Holmberg HC, Hirschberg AL, Friden C. Offered Support and Knowledge about the Menstrual Cycle in the Athletic Community: A Cross-Sectional Study of 1086 Female Athletes. Int J Environ Res Public Health. 2022 Sep 21;19(19):11932. doi: 10.3390/ijerph191911932. PMID 36231231
- [Background] Ekenros L, von Rosen P, Solli GS, Sandbakk O, Holmberg HC, Hirschberg AL, Friden C. Perceived impact of the menstrual cycle and hormonal contraceptives on physical exercise and performance in 1,086 athletes from 57 sports. Front Physiol. 2022 Aug 30;13:954760. doi: 10.3389/fphys.2022.954760. eCollection 2022. PMID 36111164
- [Background] Ekenros L, Backstrom T, Hirschberg AL, Friden C. Changes in premenstrual symptoms in women starting or discontinuing use of oral contraceptives. Gynecol Endocrinol. 2019 May;35(5):422-426. doi: 10.1080/09513590.2018.1534097. Epub 2019 Jan 22. PMID 30668208
- [Background] Von Rosen P, Kottorp A, Friden C, Frohm A, Heijne A. Young, talented and injured: Injury perceptions, experiences and consequences in adolescent elite athletes. Eur J Sport Sci. 2018 Jun;18(5):731-740. doi: 10.1080/17461391.2018.1440009. Epub 2018 Mar 3. PMID 29504456
- [Background] von Rosen P, Heijne A, Frohm A, Friden C. Menstrual irregularity and use of oral contraceptives in female adolescent athletes in Swedish National Sports High Schools. Int J Adolesc Med Health. 2017 Nov 23;32(2):/j/ijamh.2020.32.issue-2/ijamh-2017-0113/ijamh-2017-0113.xml. doi: 10.1515/ijamh-2017-0113. PMID 29168967
- [Background] Ekenros L, Papoutsi Z, Friden C, Dahlman Wright K, Linden Hirschberg A. Expression of sex steroid hormone receptors in human skeletal muscle during the menstrual cycle. Acta Physiol (Oxf). 2017 Feb;219(2):486-493. doi: 10.1111/apha.12757. Epub 2016 Aug 9. PMID 27438889
- [Background] Ekenros L, Hirschberg AL, Heijne A, Friden C. Oral contraceptives do not affect muscle strength and hop performance in active women. Clin J Sport Med. 2013 May;23(3):202-7. doi: 10.1097/JSM.0b013e3182625a51. PMID 22948447
- [Background] Ekenros L, Hirschberg AL, Backstrom T, Friden C. Postural control in women with premenstrual symptoms during oral contraceptive treatment. Acta Obstet Gynecol Scand. 2011 Jan;90(1):97-102. doi: 10.1111/j.1600-0412.2010.01021.x. Epub 2010 Nov 26. PMID 21275922
- [Background] Friden C, Ramsey DK, Backstrom T, Benoit DL, Saartok T, Linden Hirschberg A. Altered postural control during the luteal phase in women with premenstrual symptoms. Neuroendocrinology. 2005;81(3):150-7. doi: 10.1159/000086592. Epub 2005 Jun 28. PMID 15985762
- [Background] Friden C, Hirschberg AL, Saartok T, Renstrom P. Knee joint kinaesthesia and neuromuscular coordination during three phases of the menstrual cycle in moderately active women. Knee Surg Sports Traumatol Arthrosc. 2006 Apr;14(4):383-9. doi: 10.1007/s00167-005-0663-4. Epub 2005 Jun 8. PMID 15942744
- [Background] Friden C, Hirschberg AL, Saartok T, Backstrom T, Leanderson J, Renstrom P. The influence of premenstrual symptoms on postural balance and kinesthesia during the menstrual cycle. Gynecol Endocrinol. 2003 Dec;17(6):433-9. doi: 10.1080/09513590312331290358. PMID 14992161
- [Background] Friden C, Hirschberg AL, Saartok T. Muscle strength and endurance do not significantly vary across 3 phases of the menstrual cycle in moderately active premenopausal women. Clin J Sport Med. 2003 Jul;13(4):238-41. doi: 10.1097/00042752-200307000-00007. PMID 12855926
- [Background] Hirschberg AL. Challenging Aspects of Research on the Influence of the Menstrual Cycle and Oral Contraceptives on Physical Performance. Sports Med. 2022 Jul;52(7):1453-1456. doi: 10.1007/s40279-021-01616-5. Epub 2022 Jan 22. No abstract available. PMID 35064914
- [Derived] Ekenros L, von Rosen P, Norrbom J, Holmberg HC, Sundberg CJ, Friden C, Hirschberg AL. Impact of Menstrual cycle-based Periodized training on Aerobic performance, a Clinical Trial study protocol-the IMPACT study. Trials. 2024 Jan 29;25(1):93. doi: 10.1186/s13063-024-07921-4. PMID 38287424